CLINICAL TRIAL: NCT04101357
Title: Phase 1/2a, First-in-human, Open-label, Dose-escalation Trial With Expansion Cohorts to Evaluate Safety, Pharmacokinetics, Pharmacodynamics, and Preliminary Efficacy of BNT411 as a Monotherapy in Patients With Solid Tumors and in Combination With Atezolizumab, Carboplatin and Etoposide in Patients With Chemotherapy-naïve Extensive-stage Small Cell Lung Cancer (ES-SCLC)
Brief Title: Safety, Pharmacokinetics, Pharmacodynamics, and Preliminary Efficacy Trial of BNT411
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: BioNTech SE (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: BNT411-01; 2019-003593-17 (EudraCT Number)
Record Dates: First submitted 2019-09-20; First posted 2019-09-24 (Actual); Results first posted 2025-03-18 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-02

CONDITIONS: Solid Tumor; Extensive-stage Small Cell Lung Cancer
Keywords: Solid Tumor; Extensive-stage Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — atezolizumab; Carboplatin; Etoposide

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1A - monotherapy dose escalation (Experimental): BNT411 monotherapy
  Interventions: Drug: BNT411
- Part 1B - combination dose escalation (Experimental): BNT411 in combination with atezolizumab, carboplatin, and etoposide.
  Interventions: Drug: BNT411; Drug: Atezolizumab; Drug: Carboplatin; Drug: Etoposide
- Part 2 - expansion cohorts (Experimental): BNT411 either as monotherapy or in combination with atezolizumab, carboplatin, and etoposide. Please note that the sponsor decided not to continue with this part of this trial.
  Interventions: Drug: BNT411; Drug: Atezolizumab; Drug: Carboplatin; Drug: Etoposide

INTERVENTIONS:
Drug: BNT411 — intravenous
Drug: Atezolizumab — intravenous
  Arms: Part 1B - combination dose escalation; Part 2 - expansion cohorts
Drug: Carboplatin — intravenous
  Arms: Part 1B - combination dose escalation; Part 2 - expansion cohorts
Drug: Etoposide — intravenous
  Arms: Part 1B - combination dose escalation; Part 2 - expansion cohorts

SUMMARY:
This first-in-human (FIH) trial aimed to establish a safe dose of BNT411 as a monotherapy and in combination with atezolizumab, carboplatin and etoposide. BNT411 is a toll-like receptor 7 (TLR7) agonist which is expected to mount broad innate and adaptive immune reactions, especially in combination with cytotoxic therapies and immune checkpoint inhibitors.

DETAILED DESCRIPTION:
The first part (Part 1A) of this trial was a FIH, open-label, dose-escalation trial studying BNT411 monotherapy in patients with different types of malignant solid tumors in order to determine the safety profile of BNT411. The second part (Part 1B) aimed to determine further the safety profile of BNT411 in combination with atezolizumab, carboplatin and etoposide in patients with chemotherapy-naïve ES-SCLC. The third part (Part 2) was the expansion phase to explore BNT411 further as a monotherapy or in combination with atezolizumab, carboplatin and etoposide in select tumor indications. Different treatment schedules and other indications were planned to be explored in Part 2 of this trial, however, the sponsor decided not to continue with this part of this trial.

ELIGIBILITY:
Inclusion Criteria:

For Part 1A:

* Histologically confirmed solid tumor (cytology was allowed for non-small cell lung cancer [NSCLC], small cell lung cancer [SCLC] and pancreatic cancer) that was metastatic or unresectable and for which there was no available standard therapy likely to confer clinical benefit, or patients who were not candidates for such available therapy.

For Part 1B:

* Histologically or cytologically confirmed ES-SCLC (per the Veterans Administration Lung Study Group [VALG] staging system) who received no prior chemotherapy for extensive stage disease.
* Those treated with prior chemo/radiotherapy with curative intent for limited-stage small cell lung cancer (LS-SCLC) were treatment-free for at least 6 months since last chemo/radiotherapy.
* Did not have interstitial lung disease or active, non-infectious pneumonitis.

For Both Part 1A and Part 1B:

* Male and female >= 18 years of age.
* Must have signed an informed consent form (ICF) indicating that he or she understood the purpose of and procedures required for the trial and were willing to participate in the trial prior to any trial-related assessments or procedures.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
* Measurable disease according to RECIST 1.1.
* Albumin level at screening >= 30 g/L.
* Adequate coagulation function at screening as determined by:

  1. International normalized ratio (INR) or prothrombin time <= 1.5 x upper limit normal (ULN; unless on therapeutic anticoagulants with values within therapeutic window),
  2. Activated partial thromboplastin time (aPTT) <= 1.5 x ULN (unless on therapeutic anticoagulants with values within therapeutic window).
* Adequate hematologic function at screening as determined by:

  1. White blood cell count (WBC) >= 3 x 10^9/L,
  2. Absolute neutrophil count (ANC) >= 1.5 x 10^9/L (patient could not use granulocyte-colony stimulating factor (G-CSF) or granulocyte-macrophage colony stimulating factor (GM-CSF) to achieve these WBC and ANC levels),
  3. Platelet count >= 100 x 10^9/L,
  4. Hemoglobin (Hgb) >= 9.0 g/dL.
* Adequate hepatic function at screening as determined by:

  1. Total bilirubin <= 1.5 mg/dL (or <= 2.0 mg/dL for patients with known Gilbert's syndrome),
  2. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) <= 2.5 x ULN; or <= 5 x ULN in patients with metastatic liver disease.
* Adequate renal function at screening as determined by:

  a. Glomerular filtration rate (GFR) >= 60 mL/min/1.73 m^2 - e.g., according to the abbreviated Modification of Diet in Renal Disease (MDRD) equation: GFR = 186 × (SCr^-1.154) × (age^-0.203) (where SCr, the serum creatinine level, was expressed in mg/dL; multiplied by 0.742 if the patient was female; multiplied by 1.212, if the patient was African-American (Levey et al., 1999).
* Were able to attend trial visits as required by the protocol.
* Women of childbearing potential (WOCBP) must have had a negative serum (beta-human chorionic gonadotropin [beta-hCG]) test/value at screening. Patients who were postmenopausal or permanently sterilized were considered as not having reproductive potential.
* WOCBP must have agreed not to donate eggs (ova, oocytes) for the purposes of assisted reproduction during the entire trial, until 6 months after last BNT411 treatment.
* A man who was sexually active with a WOCBP and had not had a vasectomy must have agreed to use a barrier method of birth control, e.g., either condom with spermicidal foam/gel/film/cream/suppository or partner with occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository, and all men must also not donate sperm during the trial and for 6 months after receiving the last dose of BNT411.
* All patients must have provided a Formalin Fixed Paraffin Embedded (FFPE) sample from the latest available archival tumor tissue. If such tissue was not provided, the sponsor's approval of enrollment was needed.

Exclusion Criteria:

Prior and Concomitant Therapy:

* Had received prior systemic therapy with a TLR7 agonist.
* Had been receiving: radiotherapy, chemotherapy, or molecularly-targeted agents or tyrosine kinase inhibitors within 2 weeks or 5 half-lives (whichever was longer) of the start of trial treatment; immunotherapy/monoclonal antibodies within 3 weeks of the start of trial treatment; any live vaccine within 4 weeks of the start of trial treatment; nitrosoureas, antibody-drug conjugates, or radioactive isotopes within 6 weeks of the start of trial treatment.
* Received concurrent systemic (oral or intravenous) steroid therapy >10 mg prednisone daily or its equivalent for an underlying condition.
* Received concurrent strong inhibitors or inducers of the cytochrome P450 enzymes.
* Had major surgery within the 4 weeks before the first dose of BNT411.
* Had ongoing or active infection requiring intravenous treatment with anti-infective therapy that has been administered less than two weeks prior to first dose of trial treatment.
* Had side effects of any prior therapy or procedures for any medical condition not recovered to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v.5 Grade <= 1.

  * Notes: peripheral neuropathy Grade <= 2 was allowed; alopecia of any grade was allowed.

Medical Conditions

* Evidence of new or growing brain or leptomeningeal metastases during screening. Patients with known brain or leptomeningeal metastases might have been eligible if they:

  1. had radiotherapy, surgery or stereotactic surgery for the brain or leptomeningeal metastases,
  2. have no neurological symptoms (excluding Grade ≤2 neuropathy),
  3. have stable brain or leptomeningeal disease on the computed tomography (CT) or magnetic resonance imaging (MRI) scan within 4 weeks before signing the informed consent,
  4. were not undergoing acute corticosteroid therapy or steroid taper.

     * Notes: Patients with central nervous system symptoms had to undergo a CT scan or MRI of the brain to exclude new or progressive brain metastases. Spinal bone metastases were allowed, unless imminent fracture with cord compression was anticipated.
* Had history of seizures other than isolated febrile seizure in childhood; had a history of a cerebrovascular accident or transient ischemic attack less than 6 months ago.
* Had effusions (pleural, pericardial, or ascites) requiring drainage.
* Had eye pathology likely to confound observation of potential ocular adverse events.
* Had a fever >=38°C within 3 days before signing the ICF.
* Had a history of autoimmune disease active or past including but not limited to inflammatory bowel disease, systemic lupus erythematosus (SLE), ankylosing spondylitis, scleroderma, or multiple sclerosis. Had any active immunologic disorder requiring immunosuppression with steroids or other immunosuppressive agents (e.g., azathioprine, cyclosporine A) with the exception of patients with isolated vitiligo, resolved childhood asthma or atopic dermatitis, controlled hypoadrenalism or hypopituitarism, and euthyroid patients with a history of Grave's disease. Patients with controlled hyperthyroidism must have been negative for thyroglobulin, thyroid peroxidase antibodies, and thyroid-stimulating immunoglobulin prior to trial drug administration.
* Had known history of seropositivity for human immunodeficiency virus (HIV) with CD4+ T-cell (CD4+) counts <350 cells/µL and with a history of acquired immunodeficiency syndrome (AIDS)-defining opportunistic infections.
* Had known history/positive serology for hepatitis B requiring active anti-viral therapy (unless immune due to vaccination or resolved natural infection or unless passive immunization due to immunoglobulin therapy). Patients with positive serology must have had Hepatitis B virus (HBV) viral load below the limit of quantification.
* Active Hepatitis C virus (HCV) infection; patients who had completed curative antiviral treatment with HCV viral load below the limit of quantification were allowed.

  * Notes: Country-specific criteria for Germany - To confirm that a patient would be eligible, an active infection with HIV/Hepatitis B or C was ruled out by serum blood test at screening.
* Had a known hypersensitivity to a component of BNT411 drug product, or another similar compound.
* Had another primary malignancy that has not been in remission for at least 2 years, with the exception of those with a negligible risk of metastasis or death (such as adequately treated carcinoma in situ of the cervix, basal or squamous cell skin cancer, localized prostate cancer, or ductal carcinoma in situ).

Other Comorbidities

* Had abnormal electrocardiograms (ECGs) that were clinically significant, such as Framingham-corrected QT interval >480 ms.
* In the opinion of the treating investigator, had any concurrent conditions that could pose an undue medical hazard or interfere with the interpretation of the trial results; these conditions included, but were not limited to:

  1. ongoing or active infection requiring antibiotic/antiviral/antifungal therapy,
  2. concurrent congestive heart failure (New York Heart Association [NYHA] Functional Classification Class III or IV),
  3. concurrent unstable angina,
  4. concurrent cardiac arrhythmia requiring treatment (excluding asymptomatic atrial fibrillation),
  5. acute coronary syndrome within the previous 6 months,
  6. significant pulmonary disease (shortness of breath at rest or on mild exertion) for example due concurrent severe obstructive pulmonary disease.
* Had a cognitive, psychological or psychosocial impediment that would impair the ability of the patient to receive therapy according to the protocol or adversely affect the ability of the patient to comply with the informed consent process, protocol, or protocol-required visits and procedures.
* Was pregnant or breastfeeding.
* Had any contraindication to atezolizumab, carboplatin or etoposide as per US prescribing information (USPI) or summary of product characteristics (SmPC) in Part 1B.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2020-06-19 (Actual); Primary Completion 2024-01-19 (Actual); Study Completion 2024-05-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: BioNTech Responsible Person, Study Director — BioNTech SE
Locations (12):
- United States (3):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Northwestern Medical Faculty Foundation, Chicago, Illinois
  - Prisma Health-Upstate Cancer Institute, Greenville, South Carolina
- Germany (3):
  - Universitaetsklinikum Koeln - (Recruiting only for part 1B and part 2), Cologne
  - University Medical Center Hamburg-Eppendorf - (Recruiting only for part 1B and part 2), Hamburg
  - Universitaetsmedizin der Johannes Gutenberg Universitat Mainz KoeR - (Recruiting only for part 1B and part 2), Mainz
- Spain (4):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Clinica Universidad de Navarra, Madrid
  - START Madrid - CIOCC. Grupo Hospital de Madrid (HM) - Centro Integral Oncologico Clara Campal (CIOCC), Madrid
  - Hospital Universitario La Fe de Valencia, Valencia
- United Kingdom (2):
  - Edinburgh Cancer Research Centre, Edinburgh
  - Sarah Cannon Research Institute, London

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The trial was planned with three parts: Part 1A, Part 1B, and Part 2. Part 2, which was planned to consist of expansion cohorts in solid tumors was not conducted as the trial was terminated prematurely.
Groups:
- Part 1A: BNT411 Monotherapy: Dose Level (DL) 1: 0.05 mcg/kg: Participants received BNT411 at a starting dose of 0.05 micrograms per kilogram (mcg/kg) as an intravenous (IV) infusion once a week in a 3-week cycle for the first 4 cycles (on Days 1, 8, and 15; each cycle duration=21 days) followed by once every 3 weeks (on Day 1) from Cycle 5 onwards until progressive disease, unacceptable adverse events (AEs), withdrawal of consent, lost to follow-up or death whichever occurs first.
- Part 1A: BNT411 Monotherapy: DL2: 0.15 mcg/kg: Participants received BNT411 at a dose of 0.15 mcg/kg as an IV infusion once a week in a 3-week cycle for the first 4 cycles (on Days 1, 8, and 15; each cycle duration=21 days) followed by once every 3 weeks (on Day 1) from Cycle 5 onwards until progressive disease, unacceptable AE, withdrawal of consent, lost to follow-up or death whichever occurs first.
- Part 1A: BNT411 Monotherapy: DL3: 0.45 mcg/kg: Participants received BNT411 at a dose of 0.45 mcg/kg as an IV infusion once a week in a 3-week cycle for the first 4 cycles (on Days 1, 8, and 15; each cycle duration=21 days) followed by once every 3 weeks (on Day 1) from Cycle 5 onwards until progressive disease, unacceptable AE, withdrawal of consent, lost to follow-up or death whichever occurs first.
- Part 1A: BNT411 Monotherapy: DL4: 1.2 mcg/kg: Participants received BNT411 at a dose of 1.2 mcg/kg as an IV infusion once a week in a 3-week cycle for the first 4 cycles (on Days 1, 8, and 15; each cycle duration=21 days) followed by once every 3 weeks (on Day 1) from Cycle 5 onwards until progressive disease, unacceptable AE, withdrawal of consent, lost to follow-up or death whichever occurs first.
- Part 1A: BNT411 Monotherapy: DL5: 2.4 mcg/kg: Participants received BNT411 at a dose of 2.4 mcg/kg as an IV infusion once a week in a 3-week cycle for the first 4 cycles (on Days 1, 8, and 15; each cycle duration=21 days) followed by once every 3 weeks (on Day 1) from Cycle 5 onwards until progressive disease, unacceptable AE, withdrawal of consent, lost to follow-up or death whichever occurs first.
- Part 1A: BNT411 Monotherapy: DL6: 4.8 mcg/kg: Participants received BNT411 at a dose of 4.8 mcg/kg as an IV infusion once a week in a 3-week cycle for the first 4 cycles (on Days 1, 8, and 15; each cycle duration=21 days) followed by once every 3 weeks (on Day 1) from Cycle 5 onwards until progressive disease, unacceptable AE, withdrawal of consent, lost to follow-up or death whichever occurs first.
- Part 1A: BNT411 Monotherapy: DL6_2i: 6.0 mcg/kg: Participants received BNT411 at a dose of 6.0 mcg/kg as an IV infusion once a week in a 3-week cycle for the first 4 cycles (on Days 1, 8, and 15; each cycle duration=21 days) followed by once every 3 weeks (on Day 1) from Cycle 5 onwards until progressive disease, unacceptable AE, withdrawal of consent, lost to follow-up or death whichever occurs first.
- Part 1A: BNT411 Monotherapy: DL6_1i: 7.2 mcg/kg: Participants received BNT411 at a dose of 7.2 mcg/kg as an IV infusion once a week in a 3-week cycle for the first 4 cycles (on Days 1, 8, and 15; each cycle duration=21 days) followed by once every 3 weeks (on Day 1) from Cycle 5 onwards until progressive disease, unacceptable AE, withdrawal of consent, lost to follow-up or death whichever occurs first.
- Part 1A: BNT411 Monotherapy: DL7: 9.6 mcg/kg: Participants received BNT411 at a dose of 9.6 mcg/kg as an IV infusion once a week in a 3-week cycle for the first 4 cycles (on Days 1, 8, and 15; each cycle duration=21 days) followed by once every 3 weeks (on Day 1) from Cycle 5 onwards until progressive disease, unacceptable AE, withdrawal of consent, lost to follow-up or death whichever occurs first.
- Part 1B: BNT411 Combination Dose: DL4: 1.2 mcg/kg: Participants received BNT411 at a dose of 1.2 mcg/kg as an IV infusion in combination with atezolizumab, carboplatin and etoposide once a week in a 3-week cycle for the first 4 cycles (on Days 2, 8, and 15; each cycle duration=21 days) followed by once every 3 weeks (on Day 2) from Cycle 5 onwards until progressive disease, unacceptable AE, withdrawal of consent, lost to follow-up or death whichever occurs first.
- Part 1B: BNT411 Combination Dose: DL5: 2.4 mcg/kg: Participants received BNT411 at a dose of 2.4 mcg/kg as an IV infusion in combination with atezolizumab, carboplatin and etoposide once a week in a 3-week cycle for the first 4 cycles (on Days 2, 8, and 15; each cycle duration=21 days) followed by once every 3 weeks (on Day 2) from Cycle 5 onwards until progressive disease, unacceptable AE, withdrawal of consent, lost to follow-up or death whichever occurs first.
Period: Overall Study
Arm/Group | Part 1A: BNT411 Monotherapy: Dose Level (DL) 1: 0.05 mcg/kg | Part 1A: BNT411 Monotherapy: DL2: 0.15 mcg/kg | Part 1A: BNT411 Monotherapy: DL3: 0.45 mcg/kg | Part 1A: BNT411 Monotherapy: DL4: 1.2 mcg/kg | Part 1A: BNT411 Monotherapy: DL5: 2.4 mcg/kg | Part 1A: BNT411 Monotherapy: DL6: 4.8 mcg/kg | Part 1A: BNT411 Monotherapy: DL6_2i: 6.0 mcg/kg | Part 1A: BNT411 Monotherapy: DL6_1i: 7.2 mcg/kg | Part 1A: BNT411 Monotherapy: DL7: 9.6 mcg/kg | Part 1B: BNT411 Combination Dose: DL4: 1.2 mcg/kg | Part 1B: BNT411 Combination Dose: DL5: 2.4 mcg/kg
Started | 2 | 1 | 1 | 3 | 4 | 15 | 9 | 6 | 6 | 3 | 4
Safety Set (Safety set included all participants who received at least one dose of BNT411.) | 2 | 1 | 1 | 3 | 4 | 14 | 8 | 6 | 6 | 3 | 4
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 2 | 1 | 1 | 3 | 4 | 15 | 9 | 6 | 6 | 3 | 4
Not completed — Death | 1 | 1 | 1 | 2 | 4 | 11 | 4 | 4 | 5 | 2 | 3
Not completed — Trial closure | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Not completed — Other | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 0
Not completed — Enrolled but not treated | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Analysis was performed on safety set that included all participants who received at least one dose of BNT411.
Groups:
- Part 1A: BNT411 Monotherapy: DL1: 0.05 mcg/kg: Participants received BNT411 at a starting dose of 0.05 mcg/kg as an IV infusion once a week in a 3-week cycle for the first 4 cycles (on Days 1, 8, and 15; each cycle duration=21 days) followed by once every 3 weeks (on Day 1) from Cycle 5 onwards until progressive disease, unacceptable AEs, withdrawal of consent, lost to follow-up or death whichever occurs first.
- Total: Total of all reporting groups
Arm/Group | Part 1A: BNT411 Monotherapy: DL1: 0.05 mcg/kg | Part 1A: BNT411 Monotherapy: DL2: 0.15 mcg/kg | Part 1A: BNT411 Monotherapy: DL3: 0.45 mcg/kg | Part 1A: BNT411 Monotherapy: DL4: 1.2 mcg/kg | Part 1A: BNT411 Monotherapy: DL5: 2.4 mcg/kg | Part 1A: BNT411 Monotherapy: DL6: 4.8 mcg/kg | Part 1A: BNT411 Monotherapy: DL6_2i: 6.0 mcg/kg | Part 1A: BNT411 Monotherapy: DL6_1i: 7.2 mcg/kg | Part 1A: BNT411 Monotherapy: DL7: 9.6 mcg/kg | Part 1B: BNT411 Combination Dose: DL4: 1.2 mcg/kg | Part 1B: BNT411 Combination Dose: DL5: 2.4 mcg/kg | Total
Number analyzed (Participants) | 2 | 1 | 1 | 3 | 4 | 14 | 8 | 6 | 6 | 3 | 4 | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 1 | 3 | 1 | 11 | 6 | 5 | 4 | 1 | 3 | 37
  >=65 years | 1 | 0 | 0 | 0 | 3 | 3 | 2 | 1 | 2 | 2 | 1 | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 0 | 0 | 2 | 6 | 3 | 2 | 5 | 1 | 3 | 24
  Male | 1 | 0 | 1 | 3 | 2 | 8 | 5 | 4 | 1 | 2 | 1 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
  Not Hispanic or Latino | 1 | 1 | 1 | 3 | 4 | 14 | 8 | 5 | 5 | 3 | 4 | 49
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 2 | 1 | 1 | 2 | 3 | 11 | 8 | 5 | 5 | 3 | 4 | 45
  Asian | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Black or African American | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Reportable | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 1 | 0 | 0 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: DLTs were defined as any non-immune-related adverse events (AEs) or immune-related AEs during the first treatment cycle that was of Grade 3 and that did not resolve to Grade 1 or lower within a week, or that were of Grade 4. AEs were graded for severity using National Cancer Institute Common Terminology Criteria for Adverse Events, version 5.0 (NCI-CTCAE v5.0), where Grade 1: Mild; Grade 2: Moderate; Grade 3: Severe; Grade 4 - Life-threatening consequences; and Grade 5: Death related to AE.
Time Frame: Cycle 1 (21 Days)
Population: Analysis was performed on DLT evaluable set that included participants who received at least one dose of BNT411 and have completed the DLT evaluation period and meet the minimum exposure criterion or have experienced a DLT during the DLT evaluation period (Cycle 1).
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1A: BNT411 Monotherapy: DL1: 0.05 mcg/kg | Part 1A: BNT411 Monotherapy: DL2: 0.15 mcg/kg | Part 1A: BNT411 Monotherapy: DL3: 0.45 mcg/kg | Part 1A: BNT411 Monotherapy: DL4: 1.2 mcg/kg | Part 1A: BNT411 Monotherapy: DL5: 2.4 mcg/kg | Part 1A: BNT411 Monotherapy: DL6: 4.8 mcg/kg | Part 1A: BNT411 Monotherapy: DL6_2i: 6.0 mcg/kg | Part 1A: BNT411 Monotherapy: DL6_1i: 7.2 mcg/kg | Part 1A: BNT411 Monotherapy: DL7: 9.6 mcg/kg | Part 1B: BNT411 Combination Dose: DL4: 1.2 mcg/kg | Part 1B: BNT411 Combination Dose: DL5: 2.4 mcg/kg
Number analyzed (Participants) | 2 | 1 | 1 | 3 | 3 | 10 | 6 | 6 | 5 | 2 | 3
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0

2. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs), Serious TEAEs (TESAEs) and Grade >=3 TEAEs
Description: A TEAE was defined as any AE with an onset date on or after the first administration of trial treatment (if AE was absent before the first administration of trial treatment) or worsened after the first administration of trial treatment (if AE was present before the first administration of trial treatment). AEs occurring more than 60 days after last treatment administration were considered as treatment-emergent only if assessed as related to the trial treatment by the investigator. Serious adverse event (SAE): any untoward medical occurrence that, at any dose: resulted in death; was life-threatening; required inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent disability/incapacity; was a congenital anomaly/birth defect or was another medically important condition. AE were graded for severity using NCI-CTCAE v5.0, where Grade 1: Mild; Grade 2: Moderate; Grade 3: Severe; Grade 4 - Life-threatening consequences; and Grade 5: Death related to AE.
Time Frame: From Baseline until 60 days after last dose of study treatment (3 years and 11 months)
Population: Analysis was performed on safety set that included all participants who received at least one dose of BNT411.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1A: BNT411 Monotherapy: DL1: 0.05 mcg/kg | Part 1A: BNT411 Monotherapy: DL2: 0.15 mcg/kg | Part 1A: BNT411 Monotherapy: DL3: 0.45 mcg/kg | Part 1A: BNT411 Monotherapy: DL4: 1.2 mcg/kg | Part 1A: BNT411 Monotherapy: DL5: 2.4 mcg/kg | Part 1A: BNT411 Monotherapy: DL6: 4.8 mcg/kg | Part 1A: BNT411 Monotherapy: DL6_2i: 6.0 mcg/kg | Part 1A: BNT411 Monotherapy: DL6_1i: 7.2 mcg/kg | Part 1A: BNT411 Monotherapy: DL7: 9.6 mcg/kg | Part 1B: BNT411 Combination Dose: DL4: 1.2 mcg/kg | Part 1B: BNT411 Combination Dose: DL5: 2.4 mcg/kg
Number analyzed (Participants) | 2 | 1 | 1 | 3 | 4 | 14 | 8 | 6 | 6 | 3 | 4
Participants
  TEAE | 2 | 1 | 1 | 3 | 4 | 14 | 8 | 6 | 6 | 3 | 4
  Related TEAE | 2 | 1 | 0 | 2 | 1 | 13 | 7 | 6 | 6 | 3 | 4
  Grade >=3 TEAE | 1 | 0 | 1 | 0 | 3 | 3 | 3 | 5 | 5 | 3 | 3
  Related Grade >=3 TEAE | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 3 | 5 | 3 | 3
  TESAE | 1 | 0 | 1 | 0 | 1 | 5 | 3 | 4 | 3 | 2 | 3
  Related TESAE | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 3 | 3 | 2 | 2
  TESAE leading to Death | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
  Related TESAE leading to Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

3. Primary Outcome: Number of Participants Reporting Dose Reduction and/or Discontinuation of BNT411 Due to TEAEs
Description: Participants with dose reduction and/or discontinuation of BNT411 due to TEAEs are reported.
Time Frame: From Baseline until 60 days after last dose of study treatment (3 years and 11 months)
Population: Analysis was performed on safety set.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1A: BNT411 Monotherapy: DL1: 0.05 mcg/kg | Part 1A: BNT411 Monotherapy: DL2: 0.15 mcg/kg | Part 1A: BNT411 Monotherapy: DL3: 0.45 mcg/kg | Part 1A: BNT411 Monotherapy: DL4: 1.2 mcg/kg | Part 1A: BNT411 Monotherapy: DL5: 2.4 mcg/kg | Part 1A: BNT411 Monotherapy: DL6: 4.8 mcg/kg | Part 1A: BNT411 Monotherapy: DL6_2i: 6.0 mcg/kg | Part 1A: BNT411 Monotherapy: DL6_1i: 7.2 mcg/kg | Part 1A: BNT411 Monotherapy: DL7: 9.6 mcg/kg | Part 1B: BNT411 Combination Dose: DL4: 1.2 mcg/kg | Part 1B: BNT411 Combination Dose: DL5: 2.4 mcg/kg
Number analyzed (Participants) | 2 | 1 | 1 | 3 | 4 | 14 | 8 | 6 | 6 | 3 | 4
Participants
  Dose Reduction of BNT411 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 3 | 0 | 0
  Discontinuation of BNT411 due to TEAEs | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 3

4. Primary Outcome: Maximal Tolerated Dose (MTD) of BNT411
Description: The MTD defined as the highest tolerated dose was reported based on the DLTs and TEAEs experienced by participants.
Time Frame: Cycle 1 (21 days)
Population: Analysis was performed on DLT evaluable set. Data for this outcome measure was planned to be analyzed and reported for all participants collectively.
Measure: Number; unit: microgram/kilogram (mcg/kg)
Groups:
- All Participants: All Participants in Part 1A and B who received IV infusions of BNT411 every week in a 3-week cycle for the first 4 cycles (on Days 1, 8, and 15 in Part 1A; on Days 2, 8, and 15 in Part 1B; cycle duration=21 days). Thereafter, BNT411 was administered every 3 weeks (on Day 1 [Part 1A] or Day 2 [Part 1B] of each 3-week cycle) until progressive disease, unacceptable AEs, withdrawal of consent, lost to follow-up or death whichever occurs first.
Arm/Group | All Participants
Number analyzed (Participants) | 42
microgram/kilogram (mcg/kg) | 6.0

5. Primary Outcome: Recommended Phase 2 Dose (RP2D) of BNT411
Description: RP2D was based on integrated evaluation of safety, tolerability, clinical benefit, pharmacokinetic (PK), and pharmacodynamic data, for all dose levels was tested.
Time Frame: Cycle 1 (21 days)
Population: Analysis was performed on DLT evaluable population. Data for this outcome measure was planned to be analyzed and reported for all participants collectively.
Measure: Number; unit: microgram/kilogram (mcg/kg)
Arm/Group | All Participants
Number analyzed (Participants) | 42
microgram/kilogram (mcg/kg) | 4.8

6. Secondary Outcome: Pharmacokinetics (PK) Assessment for BNT411: Area Under the Concentration Time Curve (AUC0-last)
Description: AUC0-last defined as the AUC from time 0 to the last measurable time-point was calculated from plasma concentrations of BNT411 using the linear-log trapezoidal method.
Time Frame: Part 1A: Cycle 1 Day 1; Cycle 2 Day 1; Part 1B: Cycle 1 Day 2; Cycle 2 Day 2 (each cycle duration=21 days)
Population: Analysis was performed on PK evaluable set that included all participants who received at least one dose of BNT411 and have at least one quantifiable post-dose PK sample. Here, "Overall number of participants analyzed" = participants with available data for this outcome measure and number analyzed signifies participants with available data at respective visit and "0" in the number analyzed field signifies that no participants were available for analysis at the specified visit.
Measure: Mean (Standard Deviation); unit: hours (h)*picogram (pg)/milliliters (mL)
Arm/Group | Part 1A: BNT411 Monotherapy: DL1: 0.05 mcg/kg | Part 1A: BNT411 Monotherapy: DL2: 0.15 mcg/kg | Part 1A: BNT411 Monotherapy: DL3: 0.45 mcg/kg | Part 1A: BNT411 Monotherapy: DL4: 1.2 mcg/kg | Part 1A: BNT411 Monotherapy: DL5: 2.4 mcg/kg | Part 1A: BNT411 Monotherapy: DL6: 4.8 mcg/kg | Part 1A: BNT411 Monotherapy: DL6_2i: 6.0 mcg/kg | Part 1A: BNT411 Monotherapy: DL6_1i: 7.2 mcg/kg | Part 1A: BNT411 Monotherapy: DL7: 9.6 mcg/kg | Part 1B: BNT411 Combination Dose: DL4: 1.2 mcg/kg | Part 1B: BNT411 Combination Dose: DL5: 2.4 mcg/kg
Number analyzed (Participants) | 2 | 1 | 1 | 3 | 4 | 14 | 7 | 6 | 6 | 3 | 4
hours (h)*picogram (pg)/milliliters (mL)
  Cycle 1 Day 1: number analyzed (Participants) | 1 | 1 | 1 | 3 | 4 | 14 | 7 | 6 | 6 | 0 | 0
  Cycle 1 Day 1 | 187.3477 (NA) — Standard deviation could not be calculated as only 1 participant was available for the analysis. | 1477.6656 (NA) — Standard deviation could not be calculated as only 1 participant was available for the analysis. | 3123.7583 (NA) — Standard deviation could not be calculated as only 1 participant was available for the analysis. | 4724.5276 (3433.94480) | 9445.2536 (3902.75812) | 18735.9783 (11750.72661) | 22365.2916 (8763.37410) | 49384.9308 (31393.75269) | 29680.3554 (12850.18934) |  |
  Cycle 2 Day 1: number analyzed (Participants) | 2 | 1 | 1 | 3 | 3 | 10 | 3 | 4 | 4 | 0 | 0
  Cycle 2 Day 1 | 327.1261 (143.16329) | 3341.8368 (NA) — Standard deviation could not be calculated as only 1 participant was available for the analysis. | 2313.8369 (NA) — Standard deviation could not be calculated as only 1 participant was available for the analysis. | 4635.3150 (3330.49325) | 11745.1614 (2871.09499) | 20998.2267 (11223.40206) | 18392.6594 (7546.26734) | 26266.1125 (18091.16303) | 28693.3094 (7377.64393) |  |
  Cycle 1 Day 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 4
  Cycle 1 Day 2 |  |  |  |  |  |  |  |  |  | 3604.2235 (1804.20847) | 6258.0743 (1565.55574)
  Cycle 2 Day 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
  Cycle 2 Day 2 |  |  |  |  |  |  |  |  |  | 3543.6926 (4508.63205) | 3369.5271 (NA) — Standard deviation could not be calculated as only 1 participant was available for the analysis.

7. Secondary Outcome: PK Assessment for BNT411: Clearance (CL)
Description: Clearance reflects the elimination of the drug from the body was estimated from plasma concentrations of BNT411 as Dose/AUC0-inf. Dose was converted, as necessary, to reflect the amount of anhydrous BNT411 administered.
Time Frame: Part 1A: Cycle 1 Day 1; Cycle 2 Day 1; Part 1B: Cycle 1 Day 2; Cycle 2 Day 2 (each cycle duration=21 days)
Population: Analysis was performed on PK evaluable set. Here, "Overall number of participants analyzed" = participants with available data for this outcome measure and number analyzed signifies participants with available data at respective visit and "0" in the number analyzed field signifies that no participants were available for analysis at the specified visit.
Measure: Mean (Standard Deviation); unit: liters (L)/hours (h)
Groups:
- Part 1A: BNT411 Monotherapy: DL5:2.4 mcg/kg: Participants received BNT411 at a dose of 2.4 mcg/kg as an IV infusion once a week in a 3-week cycle for the first 4 cycles (on Days 1, 8, and 15; each cycle duration=21 days) followed by once every 3 weeks (on Day 1) from Cycle 5 onwards until progressive disease, unacceptable AE, withdrawal of consent, lost to follow-up or death whichever occurs first.
- Part 1B: BNT411 Combination Dose: DL5: 2.4 mcg/k: Participants received BNT411 at a dose of 2.4 mcg/kg as an IV infusion in combination with atezolizumab, carboplatin and etoposide once a week in a 3-week cycle for the first 4 cycles (on Days 2, 8, and 15; each cycle duration=21 days) followed by once every 3 weeks (on Day 2) from Cycle 5 onwards until progressive disease, unacceptable AE, withdrawal of consent, lost to follow-up or death whichever occurs first
Arm/Group | Part 1A: BNT411 Monotherapy: DL1: 0.05 mcg/kg | Part 1A: BNT411 Monotherapy: DL2: 0.15 mcg/kg | Part 1A: BNT411 Monotherapy: DL3: 0.45 mcg/kg | Part 1A: BNT411 Monotherapy: DL4: 1.2 mcg/kg | Part 1A: BNT411 Monotherapy: DL5:2.4 mcg/kg | Part 1A: BNT411 Monotherapy: DL6: 4.8 mcg/kg | Part 1A: BNT411 Monotherapy: DL6_2i: 6.0 mcg/kg | Part 1A: BNT411 Monotherapy: DL6_1i: 7.2 mcg/kg | Part 1A: BNT411 Monotherapy: DL7: 9.6 mcg/kg | Part 1B: BNT411 Combination Dose: DL4: 1.2 mcg/kg | Part 1B: BNT411 Combination Dose: DL5: 2.4 mcg/k
Number analyzed (Participants) | 1 | 1 | 1 | 3 | 4 | 14 | 7 | 5 | 6 | 2 | 4
liters (L)/hours (h)
  Cycle 1 Day 1: number analyzed (Participants) | 1 | 1 | 1 | 3 | 4 | 14 | 7 | 5 | 6 | 0 | 0
  Cycle 1 Day 1 | 27.6502 (NA) — Standard deviation could not be calculated as only 1 participant was available for the analysis. | 8.3063 (NA) — Standard deviation could not be calculated as only 1 participant was available for the analysis. | 13.1362 (NA) — Standard deviation could not be calculated as only 1 participant was available for the analysis. | 36.6351 (34.63090) | 21.1677 (8.41500) | 23.6285 (9.44317) | 24.7574 (24.89704) | 13.4479 (6.36326) | 24.4680 (9.09568) |  |
  Cycle 2 Day 1: number analyzed (Participants) | 0 | 1 | 1 | 3 | 3 | 10 | 3 | 3 | 4 | 0 | 0
  Cycle 2 Day 1 |  | 3.5213 (NA) — Standard deviation could not be calculated as only 1 participant was available for the analysis. | 17.6849 (NA) — Standard deviation could not be calculated as only 1 participant was available for the analysis. | 28.0090 (14.49788) | 13.9638 (2.28039) | 22.2684 (13.53332) | 25.7574 (14.62545) | 20.8883 (3.90723) | 21.9203 (10.72759) |  |
  Cycle 1 Day 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 4
  Cycle 1 Day 2 |  |  |  |  |  |  |  |  |  | 20.5762 (10.33093) | 30.8326 (5.92557)
  Cycle 2 Day 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Cycle 2 Day 2 |  |  |  |  |  |  |  |  |  | 14.3209 (NA) — Standard deviation could not be calculated as only 1 participant was available for the analysis. | 38.3186 (NA) — Standard deviation could not be calculated as only 1 participant was available for the analysis.

8. Secondary Outcome: PK Assessment for BNT411: Volume of Distribution (Vd)
Description: Volume of distribution (Vd) is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Vd was estimated from plasma concentrations of BNT411.
Time Frame: Part 1A: Cycle 1 Day 1; Cycle 2 Day 1; Part 1B: Cycle 1 Day 2; Cycle 2 Day 2 (each cycle duration=21 days)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: liters (L)
Arm/Group | Part 1A: BNT411 Monotherapy: DL1: 0.05 mcg/kg | Part 1A: BNT411 Monotherapy: DL2: 0.15 mcg/kg | Part 1A: BNT411 Monotherapy: DL3: 0.45 mcg/kg | Part 1A: BNT411 Monotherapy: DL4: 1.2 mcg/kg | Part 1A: BNT411 Monotherapy: DL5: 2.4 mcg/kg | Part 1A: BNT411 Monotherapy: DL6: 4.8 mcg/kg | Part 1A: BNT411 Monotherapy: DL6_2i: 6.0 mcg/kg | Part 1A: BNT411 Monotherapy: DL6_1i: 7.2 mcg/kg | Part 1A: BNT411 Monotherapy: DL7: 9.6 mcg/kg | Part 1B: BNT411 Combination Dose: DL4: 1.2 mcg/kg | Part 1B: BNT411 Combination Dose: DL5: 2.4 mcg/kg
Number analyzed (Participants) | 1 | 1 | 1 | 3 | 4 | 14 | 7 | 5 | 6 | 2 | 4
liters (L)
  Cycle 1 Day 1: number analyzed (Participants) | 1 | 1 | 1 | 3 | 4 | 14 | 7 | 5 | 6 | 0 | 0
  Cycle 1 Day 1 | 75.5414 (NA) — Standard deviation could not be calculated as only 1 participant was available for the analysis. | 47.0697 (NA) — Standard deviation could not be calculated as only 1 participant was available for the analysis. | 108.1691 (NA) — Standard deviation could not be calculated as only 1 participant was available for the analysis. | 296.6890 (313.18628) | 220.7140 (74.05373) | 232.0475 (100.19550) | 168.7668 (145.45978) | 156.7781 (77.21878) | 222.3040 (85.88236) |  |
  Cycle 2 Day 1: number analyzed (Participants) | 0 | 1 | 1 | 3 | 3 | 10 | 3 | 3 | 4 | 0 | 0
  Cycle 2 Day 1 |  | 18.6963 (NA) — Standard deviation could not be calculated as only 1 participant was available for the analysis. | 159.4620 (NA) — Standard deviation could not be calculated as only 1 participant was available for the analysis. | 194.0698 (97.37669) | 127.2646 (21.21154) | 187.7812 (96.09022) | 163.0226 (44.35908) | 186.4341 (31.41644) | 148.4863 (125.70109) |  |
  Cycle 1 Day 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 4
  Cycle 1 Day 2 |  |  |  |  |  |  |  |  |  | 132.8456 (22.90794) | 205.7365 (14.86844)
  Cycle 2 Day 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Cycle 2 Day 2 |  |  |  |  |  |  |  |  |  | 125.7815 (NA) — Standard deviation could not be calculated as only 1 participant was available for the analysis. | 243.8492 (NA) — Standard deviation could not be calculated as only 1 participant was available for the analysis.

9. Secondary Outcome: PK Assessment for BNT411: Maximum Plasma Concentration (Cmax)
Description: Cmax defined as the maximum observed plasma concentration was estimated from plasma concentrations of BNT411.
Time Frame: Part 1A: Cycle 1 Day 1; Cycle 2 Day 1; Part 1B: Cycle 1 Day 2; Cycle 2 Day 2 (each cycle duration=21 days)
Population: Analysis was performed on the PK evaluable set. Here, "Overall number of participants analyzed" = participants with available data for this outcome measure and number analyzed signifies participants with available data at respective visit and "0" in the number analyzed field signifies that no participants were available for analysis at the specified visit.
Measure: Mean (Standard Deviation); unit: picogram/milliliters (pg/mL)
Arm/Group | Part 1A: BNT411 Monotherapy: DL1: 0.05 mcg/kg | Part 1A: BNT411 Monotherapy: DL2: 0.15 mcg/kg | Part 1A: BNT411 Monotherapy: DL3: 0.45 mcg/kg | Part 1A: BNT411 Monotherapy: DL4: 1.2 mcg/kg | Part 1A: BNT411 Monotherapy: DL5: 2.4 mcg/kg | Part 1A: BNT411 Monotherapy: DL6: 4.8 mcg/kg | Part 1A: BNT411 Monotherapy: DL6_2i: 6.0 mcg/kg | Part 1A: BNT411 Monotherapy: DL6_1i: 7.2 mcg/kg | Part 1A: BNT411 Monotherapy: DL7: 9.6 mcg/kg | Part 1B: BNT411 Combination Dose: DL4: 1.2 mcg/kg | Part 1B: BNT411 Combination Dose: DL5: 2.4 mcg/kg
Number analyzed (Participants) | 2 | 1 | 1 | 3 | 4 | 14 | 7 | 6 | 6 | 3 | 4
picogram/milliliters (pg/mL)
  Cycle 1 Day 1: number analyzed (Participants) | 1 | 1 | 1 | 3 | 4 | 14 | 7 | 6 | 6 | 0 | 0
  Cycle 1 Day 1 | 152.0 (NA) — Standard deviation could not be calculated as only 1 participant was available for the analysis. | 1020.0 (NA) — Standard deviation could not be calculated as only 1 participant was available for the analysis. | 2437.0 (NA) — Standard deviation could not be calculated as only 1 participant was available for the analysis. | 3229.3 (1847.84) | 8191.3 (3211.56) | 13005.9 (4681.33) | 20404.6 (8137.20) | 31596.8 (10260.05) | 25967.7 (10270.43) |  |
  Cycle 2 Day 1: number analyzed (Participants) | 2 | 1 | 1 | 3 | 3 | 10 | 3 | 4 | 4 | 0 | 0
  Cycle 2 Day 1 | 254.0 (57.98) | 2163.0 (NA) — Standard deviation could not be calculated as only 1 participant was available for the analysis. | 1520.0 (NA) — Standard deviation could not be calculated as only 1 participant was available for the analysis. | 2947.3 (1281.14) | 8104.7 (1473.43) | 14804.4 (6042.78) | 13800.0 (3642.80) | 19551.8 (16904.30) | 22547.8 (7933.89) |  |
  Cycle 1 Day 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 4
  Cycle 1 Day 2 |  |  |  |  |  |  |  |  |  | 2880.33 (2065.462) | 5598.25 (766.713)
  Cycle 2 Day 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
  Cycle 2 Day 2 |  |  |  |  |  |  |  |  |  | 2993.95 (4214.427) | 2900.00 (NA) — Standard deviation could not be calculated as only 1 participant was available for the analysis.

10. Secondary Outcome: PK Assessment for BNT411: Time to Reach Cmax (Tmax)
Description: Tmax defined as the time to reach maximum (peak) concentration was estimated from plasma concentrations of BNT411.
Time Frame: Part 1A: Cycle 1 Day 1; Cycle 2 Day 1; Part 1B: Cycle 1 Day 2; Cycle 2 Day 2 (each cycle duration=21 days)
Population: as for outcome 9
Measure: Median (Full Range); unit: hours (h)
Arm/Group | Part 1A: BNT411 Monotherapy: DL1: 0.05 mcg/kg | Part 1A: BNT411 Monotherapy: DL2: 0.15 mcg/kg | Part 1A: BNT411 Monotherapy: DL3: 0.45 mcg/kg | Part 1A: BNT411 Monotherapy: DL4: 1.2 mcg/kg | Part 1A: BNT411 Monotherapy: DL5: 2.4 mcg/kg | Part 1A: BNT411 Monotherapy: DL6: 4.8 mcg/kg | Part 1A: BNT411 Monotherapy: DL6_2i: 6.0 mcg/kg | Part 1A: BNT411 Monotherapy: DL6_1i: 7.2 mcg/kg | Part 1A: BNT411 Monotherapy: DL7: 9.6 mcg/kg | Part 1B: BNT411 Combination Dose: DL4: 1.2 mcg/kg | Part 1B: BNT411 Combination Dose: DL5: 2.4 mcg/kg
Number analyzed (Participants) | 2 | 1 | 1 | 3 | 4 | 14 | 7 | 6 | 6 | 3 | 4
hours (h)
  Cycle 1 Day 1: number analyzed (Participants) | 1 | 1 | 1 | 3 | 4 | 14 | 7 | 6 | 6 | 0 | 0
  Cycle 1 Day 1 | 0.7667 [NA to NA] — Full range could not be calculated as only 1 participant was available for the analysis. | 0.5000 [0.500 to 0.500] | 0.5667 [NA to NA] — Full range could not be calculated as only 1 participant was available for the analysis. | 0.6500 [0.533 to 0.683] | 0.5417 [0.500 to 0.600] | 0.5917 [0.500 to 0.867] | 0.6000 [0.550 to 0.700] | 0.5417 [0.500 to 0.717] | 0.6000 [0.500 to 0.667] |  |
  Cycle 2 Day 1: number analyzed (Participants) | 2 | 1 | 1 | 3 | 3 | 10 | 3 | 4 | 4 | 0 | 0
  Cycle 2 Day 1 | 0.5750 [0.567 to 0.583] | 0.5000 [0.500 to 0.500] | 0.5833 [NA to NA] — Full range could not be calculated as only 1 participant was available for the analysis. | 0.5833 [0.583 to 0.700] | 0.5000 [0.500 to 0.583] | 0.6000 [0.500 to 0.817] | 0.6167 [0.583 to 0.617] | 0.6333 [0.567 to 0.667] | 0.6417 [0.600 to 0.750] |  |
  Cycle 1 Day 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 4
  Cycle 1 Day 2 |  |  |  |  |  |  |  |  |  | 0.5833 [0.500 to 1.017] | 0.6000 [0.500 to 0.850]
  Cycle 2 Day 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
  Cycle 2 Day 2 |  |  |  |  |  |  |  |  |  | 13.1083 [0.633 to 25.583] | 0.5833 [NA to NA] — Full range could not be calculated as only 1 participant was available for the analysis.

11. Secondary Outcome: PK Assessment for BNT411: Trough Concentration (Ctrough)
Description: Ctrough defined as the pre-dose concentrations of BNT411 was estimated from the plasma concentrations of BNT411.
Time Frame: Part 1A: Start of infusion on Cycle 1 Day 8, Day 15, Day 22, Day 43; Day 85; Part 1B: Start of infusion on Cycle 1 Day 8, Day 15, Day 23, Day 44 (each cycle duration=21 days)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: picogram/milliliters (pg/mL)
Arm/Group | Part 1A: BNT411 Monotherapy: DL1: 0.05 mcg/kg | Part 1A: BNT411 Monotherapy: DL2: 0.15 mcg/kg | Part 1A: BNT411 Monotherapy: DL3: 0.45 mcg/kg | Part 1A: BNT411 Monotherapy: DL4: 1.2 mcg/kg | Part 1A: BNT411 Monotherapy: DL5: 2.4 mcg/kg | Part 1A: BNT411 Monotherapy: DL6: 4.8 mcg/kg | Part 1A: BNT411 Monotherapy: DL6_2i: 6.0 mcg/kg | Part 1A: BNT411 Monotherapy: DL6_1i: 7.2 mcg/kg | Part 1A: BNT411 Monotherapy: DL7: 9.6 mcg/kg | Part 1B: BNT411 Combination Dose: DL4: 1.2 mcg/kg | Part 1B: BNT411 Combination Dose: DL5: 2.4 mcg/kg
Number analyzed (Participants) | 2 | 1 | 1 | 3 | 4 | 8 | 6 | 2 | 4 | 2 | 4
picogram/milliliters (pg/mL)
  Cycle 1 Day 8: number analyzed (Participants) | 1 | 1 | 1 | 2 | 1 | 8 | 6 | 2 | 4 | 2 | 1
  Cycle 1 Day 8 | 0.000 (NA) — Standard deviation could not be calculated as only 1 participant was available for the analysis. | 0.000 (NA) — Standard deviation could not be calculated as only 1 participant was available for the analysis. | 0.000 (NA) — Standard deviation could not be calculated as only 1 participant was available for the analysis. | 0.000 (0.0000) | 0.000 (NA) — Standard deviation could not be calculated as only 1 participant was available for the analysis. | 0.476 (0.9789) | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000) | 0.0 (0.00) | 0.0 (NA) — Standard deviation could not be calculated as only 1 participant was available for the analysis.
  Cycle 1 Day 15: number analyzed (Participants) | 2 | 0 | 1 | 3 | 4 | 6 | 4 | 2 | 2 | 1 | 4
  Cycle 1 Day 15 | 8.400 (11.8794) |  | 0.000 (NA) — Standard deviation could not be calculated as only 1 participant was available for the analysis. | 0.000 (0.0000) | 0.253 (0.5050) | 0.168 (0.4123) | 0.580 (0.6722) | 1.350 (0.2970) | 1.655 (0.5303) | 0.0 (NA) — Standard deviation could not be calculated as only 1 participant was available for the analysis. | 0.0 (0.00)
  Cycle 1 Day 22: number analyzed (Participants) | 2 | 0 | 1 | 2 | 2 | 8 | 2 | 1 | 1 | 0 | 0
  Cycle 1 Day 22 | 0.000 (0.0000) |  | 0.000 (NA) — Standard deviation could not be calculated as only 1 participant was available for the analysis. | 51.500 (72.8320) | 0.000 (0.0000) | 0.000 (0.0000) | 0.000 (0.0000) | 1.770 (NA) — Standard deviation could not be calculated as only 1 participant was available for the analysis. | 0.000 (NA) — Standard deviation could not be calculated as only 1 participant was available for the analysis. |  |
  Cycle 1 Day 23: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Cycle 1 Day 23 |  |  |  |  |  |  |  |  |  |  | 0.0 (NA) — Standard deviation could not be calculated as only 1 participant was available for the analysis.
  Cycle 1 Day 43: number analyzed (Participants) | 1 | 0 | 0 | 3 | 1 | 3 | 1 | 2 | 1 | 0 | 0
  Cycle 1 Day 43 | 0.000 (NA) — Standard deviation could not be calculated as only 1 participant was available for the analysis. |  |  | 4.833 (8.3716) | 0.000 (NA) — Standard deviation could not be calculated as only 1 participant was available for the analysis. | 0.370 (0.6409) | 0.000 (NA) — Standard deviation could not be calculated as only 1 participant was available for the analysis. | 0.970 (1.3718) | 1.690 (NA) — Standard deviation could not be calculated as only 1 participant was available for the analysis. |  |
  Cycle 1 Day 44: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Cycle 1 Day 44 |  |  |  |  |  |  |  |  |  | 0.0 (NA) — Standard deviation could not be calculated as only 1 participant was available for the analysis. | 0.0 (NA) — Standard deviation could not be calculated as only 1 participant was available for the analysis.
  Cycle 1 Day 85: number analyzed (Participants) | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 1 | 0 | 0
  Cycle 1 Day 85 |  |  |  | 0.590 (0.8344) |  |  | 38500.000 (NA) — Standard deviation could not be calculated as only 1 participant was available for the analysis. | 1.170 (NA) — Standard deviation could not be calculated as only 1 participant was available for the analysis. | 0.000 (NA) — Standard deviation could not be calculated as only 1 participant was available for the analysis. |  |

12. Secondary Outcome: PK Assessment for BNT411: Terminal Elimination Half-life (T1/2)
Description: Terminal elimination half-life was estimated from the plasma concentrations of BNT411.
Time Frame: Part 1A: Cycle 1 Day 1; Cycle 2 Day 1; Part 1B: Cycle 1 Day 2; Cycle 2 Day 2 (each cycle duration=21 days)
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: hours (h)
Arm/Group | Part 1A: BNT411 Monotherapy: DL1: 0.05 mcg/kg | Part 1A: BNT411 Monotherapy: DL2: 0.15 mcg/kg | Part 1A: BNT411 Monotherapy: DL3: 0.45 mcg/kg | Part 1A: BNT411 Monotherapy: DL4: 1.2 mcg/kg | Part 1A: BNT411 Monotherapy: DL5: 2.4 mcg/kg | Part 1A: BNT411 Monotherapy: DL6: 4.8 mcg/kg | Part 1A: BNT411 Monotherapy: DL6_2i: 6.0 mcg/kg | Part 1A: BNT411 Monotherapy: DL6_1i: 7.2 mcg/kg | Part 1A: BNT411 Monotherapy: DL7: 9.6 mcg/kg | Part 1B: BNT411 Combination Dose: DL4: 1.2 mcg/kg | Part 1B: BNT411 Combination Dose: DL5: 2.4 mcg/kg
Number analyzed (Participants) | 1 | 1 | 1 | 3 | 4 | 14 | 7 | 5 | 6 | 2 | 4
hours (h)
  Cycle 1 Day 1: number analyzed (Participants) | 1 | 1 | 1 | 3 | 4 | 14 | 7 | 5 | 6 | 0 | 0
  Cycle 1 Day 1 | 1.8937 (NA) — Standard deviation could not be calculated as only 1 participant was available for the analysis. | 3.9279 (NA) — Standard deviation could not be calculated as only 1 participant was available for the analysis. | 5.7077 (NA) — Standard deviation could not be calculated as only 1 participant was available for the analysis. | 5.2525 (0.99582) | 7.4679 (1.87347) | 7.4600 (4.30673) | 5.1189 (1.23014) | 8.7346 (4.71577) | 6.2721 (0.48131) |  |
  Cycle 2 Day 1: number analyzed (Participants) | 0 | 1 | 1 | 3 | 3 | 10 | 3 | 3 | 4 | 0 | 0
  Cycle 2 Day 1 |  | 3.6803 (NA) — Standard deviation could not be calculated as only 1 participant was available for the analysis. | 6.2500 (NA) — Standard deviation could not be calculated as only 1 participant was available for the analysis. | 4.9020 (0.57744) | 6.3386 (0.73577) | 6.0603 (1.18916) | 4.9479 (1.51079) | 6.2166 (0.45957) | 4.5667 (2.07892) |  |
  Cycle 1 Day 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 4
  Cycle 1 Day 2 |  |  |  |  |  |  |  |  |  | 4.8989 (1.68795) | 4.7244 (0.68988)
  Cycle 2 Day 2: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Cycle 2 Day 2 |  |  |  |  |  |  |  |  |  | 6.0880 (NA) — Standard deviation could not be calculated as only 1 participant was available for the analysis. | 4.4110 (NA) — Standard deviation could not be calculated as only 1 participant was available for the analysis.

ADVERSE EVENTS:
Time Frame: From Baseline until 60 days after the last dose of study treatment (3 years and 11 months)
Description: All-cause mortality analysis was performed on all enrolled participants. All SAEs and Non-Serious AEs data collected through-out the study are reported in the AE section and analysis was performed on safety analysis set (that is, all participants who received at least one dose of BNT411).
Groups:
- Part 1A: BNT411 Monotherapy: Dose Level (DL) 1: 0.05 mcg/kg: Participants received BNT411 at a starting dose of 0.05 mcg/kg as an IV infusion once a week in a 3-week cycle for the first 4 cycles (on Days 1, 8, and 15; each cycle duration=21 days) followed by once every 3 weeks (on Day 1) from Cycle 5 onwards until progressive disease, unacceptable AEs, withdrawal of consent, lost to follow-up or death whichever occurs first.
Arm/Group | Part 1A: BNT411 Monotherapy: Dose Level (DL) 1: 0.05 mcg/kg | Part 1A: BNT411 Monotherapy: DL2: 0.15 mcg/kg | Part 1A: BNT411 Monotherapy: DL3: 0.45 mcg/kg | Part 1A: BNT411 Monotherapy: DL4: 1.2 mcg/kg | Part 1A: BNT411 Monotherapy: DL5: 2.4 mcg/kg | Part 1A: BNT411 Monotherapy: DL6: 4.8 mcg/kg | Part 1A: BNT411 Monotherapy: DL6_2i: 6.0 mcg/kg | Part 1A: BNT411 Monotherapy: DL6_1i: 7.2 mcg/kg | Part 1A: BNT411 Monotherapy: DL7: 9.6 mcg/kg | Part 1B: BNT411 Combination Dose: DL4: 1.2 mcg/kg | Part 1B: BNT411 Combination Dose: DL5: 2.4 mcg/kg
All-Cause Mortality (participants affected / at risk) | 1/2 | 1/1 | 1/1 | 2/3 | 4/4 | 11/15 | 4/9 | 4/6 | 5/6 | 2/3 | 3/4
Serious Adverse Events (participants affected / at risk) | 1/2 | 0/1 | 1/1 | 1/3 | 1/4 | 5/14 | 3/8 | 4/6 | 4/6 | 2/3 | 3/4
Other Adverse Events (participants affected / at risk) | 2/2 | 1/1 | 1/1 | 3/3 | 4/4 | 14/14 | 8/8 | 6/6 | 6/6 | 3/3 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1A: BNT411 Monotherapy: Dose Level (DL) 1: 0.05 mcg/kg (N=2) | Part 1A: BNT411 Monotherapy: DL2: 0.15 mcg/kg (N=1) | Part 1A: BNT411 Monotherapy: DL3: 0.45 mcg/kg (N=1) | Part 1A: BNT411 Monotherapy: DL4: 1.2 mcg/kg (N=3) | Part 1A: BNT411 Monotherapy: DL5: 2.4 mcg/kg (N=4) | Part 1A: BNT411 Monotherapy: DL6: 4.8 mcg/kg (N=14) | Part 1A: BNT411 Monotherapy: DL6_2i: 6.0 mcg/kg (N=8) | Part 1A: BNT411 Monotherapy: DL6_1i: 7.2 mcg/kg (N=6) | Part 1A: BNT411 Monotherapy: DL7: 9.6 mcg/kg (N=6) | Part 1B: BNT411 Combination Dose: DL4: 1.2 mcg/kg (N=3) | Part 1B: BNT411 Combination Dose: DL5: 2.4 mcg/kg (N=4)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Diplopia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Disease progression (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 3 | 2 | 0 | 1
COVID-19 (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Device related infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Tumour thrombosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Dysarthria (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Immune effector cell-associated neurotoxicity syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Mental status changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Superior vena cava syndrome (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1A: BNT411 Monotherapy: Dose Level (DL) 1: 0.05 mcg/kg (N=2) | Part 1A: BNT411 Monotherapy: DL2: 0.15 mcg/kg (N=1) | Part 1A: BNT411 Monotherapy: DL3: 0.45 mcg/kg (N=1) | Part 1A: BNT411 Monotherapy: DL4: 1.2 mcg/kg (N=3) | Part 1A: BNT411 Monotherapy: DL5: 2.4 mcg/kg (N=4) | Part 1A: BNT411 Monotherapy: DL6: 4.8 mcg/kg (N=14) | Part 1A: BNT411 Monotherapy: DL6_2i: 6.0 mcg/kg (N=8) | Part 1A: BNT411 Monotherapy: DL6_1i: 7.2 mcg/kg (N=6) | Part 1A: BNT411 Monotherapy: DL7: 9.6 mcg/kg (N=6) | Part 1B: BNT411 Combination Dose: DL4: 1.2 mcg/kg (N=3) | Part 1B: BNT411 Combination Dose: DL5: 2.4 mcg/kg (N=4)
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 2 | 1 | 1 | 1 | 3 | 3 | 2 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Atrioventricular block first degree (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Myopericarditis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blepharitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Eye irritation (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Eye pruritus (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Meibomian gland dysfunction (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Retinal exudates (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Retinal haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Visual field defect (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Visual impairment (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vitreous detachment (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 5 | 1 | 0 | 1 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 2 | 1 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lip dry (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 8 | 3 | 2 | 5 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0 | 3 | 2 | 3 | 5 | 0 | 0
Asthenia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 0
Axillary pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 1 | 0 | 0 | 0 | 0 | 2 | 2 | 3 | 4 | 0 | 0
Energy increased (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Face oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 1 | 2 | 6 | 3 | 3 | 5 | 1 | 0
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
General physical health deterioration (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Generalised oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 1 | 0 | 0 | 1 | 5 | 3 | 3 | 2 | 1 | 1
Hepatic pain (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cytokine release syndrome (Immune system disorders) | 0 | 0 | 0 | 1 | 0 | 3 | 5 | 3 | 4 | 0 | 0
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
COVID-19 (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Herpes simplex reactivation (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oesophageal candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 3 | 0 | 1 | 0 | 0 | 0
Joint injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 2 | 0 | 0
Amylase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 2 | 3 | 0 | 2 | 1 | 0
Bacterial test positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 2 | 1 | 0 | 0
Blood calcium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 2
Blood fibrinogen decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0
Blood potassium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood potassium increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood thyroid stimulating hormone increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
C-reactive protein increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
International normalised ratio increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Liver function test increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 3 | 1 | 2 | 1
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 2 | 2
Respiratory rate increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Troponin I increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0
Weight increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1
White blood cells urine positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 3 | 3 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 2 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 1 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 3 | 3 | 0 | 0
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0
Brain fog (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 3 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 1 | 0 | 3 | 2 | 2 | 3 | 0 | 0
Hemiparesis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Neurotoxicity (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 1 | 0 | 0
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Sleep disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Social avoidant behaviour (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Chromaturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 0 | 0
Micturition urgency (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nocturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oliguria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 2 | 1 | 2 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 1 | 2 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2 | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Embolism (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 1 | 0 | 0
Hypotension (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 3 | 0 | 1 | 1 | 0 | 0

LIMITATIONS AND CAVEATS:
The planned Part 2 of the study was not conducted as the trial was terminated prematurely.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigators respectively trial sites shall not publish or refer to in writing or orally, in whole or in part, any data, information or materials generated from the study and the services, without the prior written consent of the sponsor.

DOCUMENTS (2):
  • Study Protocol (2023-07-04): https://cdn.clinicaltrials.gov/large-docs/57/NCT04101357/Prot_000.pdf
  • Statistical Analysis Plan (2024-02-21): https://cdn.clinicaltrials.gov/large-docs/57/NCT04101357/SAP_001.pdf